CLINICAL TRIAL: NCT05686096
Title: A Phase 1, Open-label, Single Dose Study to Assess the Absorption, Metabolism, and Excretion of [14C]BMS-986435 in Healthy Male Participants
Brief Title: A Study to Evaluate the Absorption, Metabolism, and Excretion (ADME) of BMS-986435
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV029-012
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
Keywords: Absorption, Metabolism, and Excretion (ADME); MYK-224

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MYK-224 (Experimental)
  Interventions: Drug: MYK-224

INTERVENTIONS:
Drug: MYK-224 — Specified dose on specified days
  Other Names: BMS-986435

SUMMARY:
The purpose of this study is to determine the absorption, metabolism, excretion; and to evaluate the safety and tolerability of BMS-986435 in healthy male participants

Participants will be admitted to the study site for 3 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index between 18 and 32 kg/m^2, inclusive, at screening. - Healthy male participants as determined by the investigator and sponsor.
* Adequate acoustic windows to enable accurate transthoracic echocardiogram (TTE) assessment of parameters of left ventricular (LV) systolic function by TTE.
* Documented left ventricular ejection fraction (LVEF) ≥ 60% at screening.

Key Exclusion Criteria:

* Any acute or chronic medical illness.
* History of dizziness and/or recurrent headaches (ie, daily headaches lasting for a 1-week duration in the last month prior to study intervention administration).

Head injury in the last 2 years, intracranial tumor, or aneurysm. Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-04-08 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 45 days
Time to maximum observed concentration (Tmax) | Up to 45 days
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Up to 45 days

SECONDARY OUTCOMES:
Metabolite profiling of BMS-986435 in plasma, urine, and feces | Up to 45 days
Number of participants with adverse events (AEs) | Up to 45 days
Number of participants with clinical laboratory abnormalities | Up to 45 days
Number of participants with vital sign abnormalities | Up to 45 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 45 days
Number of participants with physical examination abnormalities | Up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol-Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.htm

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm